CLINICAL TRIAL: NCT02811874
Title: Efficacy of Community Health Workers Education in Diabetes Control: A Randomized Clinical Trial
Brief Title: Community Health Workers and Diabetes Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09-069
Record Dates: First submitted 2016-03-04; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes
Keywords: diabetes education; community health workers; diabetes control
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- diabetes education (Experimental): Four community health workers receive a one-month diabetes education program (intervention group, patients n= 62)
  Interventions: Behavioral: diabetes education
- education in other areas (Active Comparator): Four community health workers receive an education course in other health issues (control group, patients n= 56).
  Interventions: Behavioral: education in other areas

INTERVENTIONS:
Behavioral: diabetes education — Diabetes education program includes: 4 theoretical sessions, 60 minutes long, taught once a week for 4 weeks, developed in the form of group classes, and given by one of the authors. The educational program content comprises (1) definition of diabetes, and identification of modifiable risk factors for type 2 diabetes, (2) non-pharmacological treatment, with emphasis on diet and exercise, (3) pharmacological therapy, including mechanism of action and side effects of anti-diabetic medications provided by the Brazilian public health system and (4) an overview of chronic diabetes complications.
  Arms: diabetes education
Behavioral: education in other areas — Four theoretical sessions related to education in other health areas, not related to diabetes, administered during 4 weeks
  Arms: education in other areas

SUMMARY:
The aim of this study is to evaluate the effect of a diabetes education program delivered to CHW in improving the metabolic control of patients with type 2 DM.

The study is a randomized controlled trial conducted in a primary care unit. Eight CHW, providing care for 118 patients, are randomized in two groups to receive a one-month diabetes education program (intervention group, patients n= 62) or an education course in other health issues (control group, patients n= 56).

DETAILED DESCRIPTION:
Background: In Brazil, community health workers (CHW) are members of the community hired by the government to provide education and care for patients for a broad range of health issues, including diabetes mellitus (DM). However, few CHW are trained for diabetes education and little is known about the effectiveness of their interventions. The aim of this study is to evaluate the effect of a diabetes education program delivered to CHW in improving the metabolic control of patients with type 2 DM.

Materials and methods: the study is a randomized controlled trial conducted in a primary care unit. Eight CHW, providing care for 118 patients, are randomized in two groups to receive a one-month diabetes education program (intervention group, patients n= 62) or an education course in other health issues (control group, patients n= 56). Each CHW is responsible for transmitting the acquired knowledge to patients from their respective working areas. The primary outcome is change in HbA1C three months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with diabetes mellitus who live in the community of the health care unit and who agree to participate the study.

Exclusion Criteria:

* None.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | comparison baseline and three months after intervention.

SECONDARY OUTCOMES:
Diabetes literacy | comparison baseline and three months after intervention.
  measured by a 22 questions questionnaire testing diabetes knowledge
Diastolic Blood pressure | comparison baseline and three months after intervention.
  unit: mmHg
Systolic Blood Pressure | comparison baseline and three months after intervention.
  unit: mmHg
Total cholesterol | comparison baseline and three months after intervention.
  unit: mg/dL
HDL-Cholesterol | comparison baseline and three months after intervention.
  unit: mg/dL
Triglycerides | comparison baseline and three months after intervention.
  unit: mg/dL
Height | baseline measure only
  unit: centimeters; this outcome will be used to calculate Body Mass Index (BMI)
Weight | comparison baseline and three months after intervention.
  unit: kilograms; this outcome will be used to calculate Body Mass Index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Bauermann Leitão, PhD, Study Director — HCPA/UFRGS
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UBS São Pedro, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided